CLINICAL TRIAL: NCT02497976
Title: Pilot Study Evaluating the Efficacy of Certolizumab Pegol for Interstitial Cystitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ICStudy, LLC (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Philip C. Bosch, M.D., Philip C Bosch, MD, ICStudy, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IC-201
Record Dates: First submitted 2015-07-10; First posted 2015-07-15 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Cystitis, Interstitial
Keywords: Interstitial; Cystitis; Bladder; Pain
MeSH Terms: conditions — Cystitis, Interstitial; Cystitis; Pain | interventions — Certolizumab Pegol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Experimental (Active Comparator): Biological: Certolizumab pegol (Cimzia) 400 mg loading dose given subcutaneously at week 0, 2, and 4 followed by a maintenance dose at week 8
  Interventions: Biological: Certolizumab pegol
- Group 2: Placebo Comparator (Placebo Comparator): Placebo: given subcutaneously at week 0, 2, 4, and week 8
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Certolizumab pegol — 400 mg
  Other Names: Cimzia
  Arms: Group 1: Experimental
Drug: Placebo — Normal saline
  Other Names: Normal saline
  Arms: Group 2: Placebo Comparator

SUMMARY:
A Randomized, Double-blind, Placebo Controlled Trial of Certolizumab Pegol in Women with Refractory Interstitial Cystitis/Bladder Pain Syndrome

DETAILED DESCRIPTION:
Interstitial cystitis (IC) is a chronic disabling bladder syndrome characterized by urinary frequency, nocturia, urinary urgency, and pain or discomfort with bladder filling. There is no cure for IC and the treatment options are suboptimal. Patients with IC report significant negative effects on their physical and mental quality of life. The etiology of IC is unknown. Certain aspects of IC suggest that autoimmunity may play a role in initiating or sustaining the chronic inflammatory response. Bladder biopsies of patients with IC demonstrate an increase number of mast cells. Mast cell activation with the release of tumor necrosis factor (TNF) may mediate this bladder inflammation. Cimzia (certolizumab pegol) is a medication that blocks the effect of TNF. Cimzia (certolizumab pegol) is FDA approved for the treatment of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, and Crohn's disease. These diseases are similar to IC. In this study, the hypothesis being tested is that Cimzia (certolizumab pegol) will show efficacy in improving the symptoms of patients with IC.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of IC/BPS defined based on AUA guidelines as the following: an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than 6 months duration, in the absence of infection or identifiable causes, documented history or patient reported.
2. Only those patients with moderate to severe IC/BPS will be included in the study.
3. Able to provide informed consent to participate in the study and comply with study requirements
4. Able to provide written authorization for use and release of health and research study information
5. Written documentation of being provided California's Experimental Subject's Bill of Rights
6. Females ≥18 and ≤ 65 years of age previously diagnosed with interstitial cystitis/ bladder pain syndrome (IC/BPS) for a duration of greater than 6 months
7. Female patients of child-bearing potential must have a negative serum pregnancy test at Screening and use birth control while in the study.
8. O'Leary-Sant Interstitial Cystitis Symptom and Problem Indexes (OSPI) score ≥ 18
9. No history of any cancer.
10. No bacterial cystitis in previous 1 month
11. No active herpes in previous 3 months
12. Never treated with cyclophosphamide
13. No neurogenic bladder dysfunction (due to a spinal cord injury, stroke, Parkinson's disease, multiple sclerosis, spina bifida or diabetic cystopathy)
14. Absence of bladder, ureteral or urethral calculi for previous 3 months

Exclusion criteria:

1. Symptoms are relieved at one month reevaluation visit after receiving IC/BPS behavior modification advice at screening visit.
2. Symptoms are relieved by antimicrobials, antibiotics, or other medications for IC/BPS
3. Pregnant women, lactating mothers, nursing mothers, women suspected of being pregnant and woman who plan to be pregnant during the course of the clinical trial
4. Males
5. Patients with inadequate renal, hepatic, or cardiac function
6. Patients with history of gross hematuria within 2 years.
7. Patients with the following medical history: Lower urinary tract anatomical anomaly, pelvic radiotherapy, or active genital herpes
8. Patients with a history of tuberculosis (TB), recent exposure to TB, or recent travel to TB endemic regions. Patients should have a recent negative PPD (or negative CXR) prior to receiving treatment.
9. Patients who have undergone cystoscopy under anesthesia with bladder biopsy, hydrodistension, or fulguration of Hunner's ulcer within 3 months
10. Patients taking the following treatments for interstitial cystitis at Screening: Intravesical BCG, corticosteroid therapy, cyclosporine, or TNF-alpha inhibitors.
11. Patients with a history of receiving live vaccine including Flumist® influenza vaccine in the past 3 months.
12. Patients with a history of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG-fusion protein.
13. Patients with a history of alcohol, analgesic or drug abuse within 2 years of Screening.
14. Patients with a history of any cancer.
15. Patients with a history of active Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV) infection, or who are known carriers (Hepatitis B).
16. Patients with a history of invasive fungal infections, recent travel to regions endemic for the following invasive fungal infections: San Joaquin Fever, aspergillosis, histoplasmosis, candidiasis, coccidiodomycosis, blastomycosis, and pneumocystosis.
17. Patients with a history of diabetes mellitus.
18. Patients with a history of a neurologic disease included but not limited to central demyelinating diseases, including multiple sclerosis; and a history of peripheral demyelinating disease, including Guillain-Barre syndrome.
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-04-16 (Actual); Study Completion 2017-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Bosch, MD, Principal Investigator — IC Study, LLC
Locations (1):
- Philip C. Bosch, MD, Escondido, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosch PC. A randomized, double-blind, placebo controlled trial of adalimumab for interstitial cystitis/bladder pain syndrome. J Urol. 2014 Jan;191(1):77-82. doi: 10.1016/j.juro.2013.06.038. Epub 2013 Jun 20. PMID 23792149
- [Result] Bosch PC. Examination of the significant placebo effect in the treatment of interstitial cystitis/bladder pain syndrome. Urology. 2014 Aug;84(2):321-6. doi: 10.1016/j.urology.2014.04.011. Epub 2014 Jun 21. PMID 24958479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from my practice, web site, and Urology clinic at UCSD from December 10, 2015 through March 1, 2017.
Pre-assignment Details: There were 3 patients who did not meet screening criteria. Twenty-four patients had sufficient improvement in their IC/BPS symptoms and did not continue with the drug versus placebo phase of the study.
Period: Overall Study
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
Started | 28 | 14
Completed | 26 | 13
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Moved out of area | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Certolizumab Pegol: Experimental drug certolizumab pegol 400mg.
- Total: Total of all reporting groups
Arm/Group | Certolizumab Pegol | Placebo | Total
Number analyzed (Participants) | 28 | 14 | 42
Age, Continuous [Median (Standard Deviation); unit: years] | 46.9 (12.7) | 49.9 (10.7) | 47.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Only females between the age of 18 to 65.
  Participants
    Female | 28 | 14 | 42
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 24 | 13 | 37
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Count of participants]
  United States | 28 | 14 | 42
O'Leary Sant Symptom and Problem Index [Mean (Standard Deviation); unit: units on a scale] — Subjects rated the presence and extent of IC/BPS symptoms by completing the O'Leary-Sant Interstitial Cystitis Symptom Index and the O'Leary-Sant Interstitial Cystitis Problem Index (ICPI) at baseline and at weeks 2, 4, 10, and 18. Lubeck et al validated ICSI as a valid measure of change in treatment outcome studies. Propert et al validated the ICSI as responsive to change in IC/BPS symptoms and was recommended as secondary endpoints in clinical trials. No urinary symptoms would have a score of 0. The most severe symptoms would be a maximum of 35. Normal patients have a value of 7 or less.
  units on a scale | 26.8 (5.2) | 26.7 (4.8) | 26.8 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: IC/BPS Symptoms Change With Overall Global Response Assessment (GRA)
Description: Patient-reported global response assessment (GRA) such as "Compared to when you began this trial, how would you rate your IC symptoms now?" Study subjects reported their response to treatment of their pain, urgency, and overall status compared to their condition at trial start with a symmetric scale global response assessment (GRA) 28 at weeks 2, 4, 10, and 18. Possible responses were markedly worse (100% worse), moderately worse (50% worse), slightly worse (25% worse), no change (0% improvement), slightly improved (25% improvement), moderately improved (50% improvement), and markedly improved (100% improved). Treatment responders were defined by rating the GRA as moderately improved or markedly improved.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
Number analyzed (Participants) | 28 | 14
Participants | 2 | 1

2. Secondary Outcome: IC/BPS Symptoms Change With Overall Global Response Assessment (GRA)
Description: as for outcome 1
Time Frame: Week 4, 10, 18
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
Number analyzed (Participants) | 28 | 14
Participants
  Week 4 | 8 | 3
  Week 10 | 12 | 3
  Week 18 | 15 | 1

3. Secondary Outcome: IC/BPS Symptoms Assessment With the Interstitial Cystitis Symptom Index
Description: The Interstitial Cystitis Symptom Index is one of the two O'Leary-Sant Interstitial Cystitis Symptom and Problem Indexes. This scale has a 0 if the patient has no symptoms and a maximum of 19 with severe symptoms. Lubeck et al. validated ICSI as a valid measure of change in treatment outcome studies. A change of -4.03 in the ICSI score was the same as a 2 point improvement in GRA. Propert et al. validated the ICSI as responsive to change in IC/BPS symptoms and was recommended as secondary endpoints in clinical trials. A change of -2.4 in the ICSI score was the same as a 2 point improvement in GRA.
Time Frame: Value at Weeks 2, 4, 10 and 18 minus Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
Number analyzed (Participants) | 28 | 14
units on a scale
  Week 2 | -1.9 (2.7) | -0.6 (2.4)
  Week 4 | -3.3 (3.4) | -1.5 (3.0)
  Week 10 | -4.1 (4.8) | -2.8 (3.2)
  Week 18 | -5.1 (4.9) | -1.5 (4.6)

4. Secondary Outcome: IC/BPS Symptoms Assessment With the Interstitial Cystitis Problem Index (ICPI)
Description: The Interstitial Cystitis Symptom Index (ICPI) is one of the two O'Leary-Sant Interstitial Cystitis Symptom and Problem Indexes. This scale has a 0 if the patient has no symptoms and a maximum of 16 with severe symptoms.
Time Frame: Value of Weeks 2, 4, 10, and 18 minus baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
Number analyzed (Participants) | 28 | 14
units on a scale
  Week 2 | -1.4 (2.4) | -1.4 (2.0)
  Week 4 | -2.3 (3.4) | -2.3 (4.0)
  Week 10 | -4.1 (4.4) | -2.3 (3.2)
  Week 18 | -4.8 (4.8) | -1.8 (3.9)

5. Secondary Outcome: Pain Scale
Description: an 11-point pain intensity numerical rating scale. Subjects rated their average pain, pressure, or discomfort associated with their bladder using an 11-point pain intensity numerical rating scale of 0-no pain to 10-worse ever pain at baseline, and at weeks 2, 4, 10, and 18. Meaningful, clinically important pain relief is a reduction in pain of approximately 30% from baseline.
Time Frame: Value at Weeks 2, 4, 10, and 18 minus baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
Number analyzed (Participants) | 28 | 14
units on a scale
  Week 2 | -0.9 (1.7) | -0.8 (1.8)
  Week 4 | -1.1 (1.9) | -0.1 (1.4)
  Week 10 | -2.0 (2.8) | -0.6 (2.1)
  Week 18 | -2.4 (2.9) | -0.4 (2.2)

6. Secondary Outcome: Urgency Scale
Description: Subjects rated their average urinary urgency or need to urinate using an 11-point numerical rating scale of 0-no urgency to 10-worse ever urgency
Time Frame: Value of Weeks 2, 4, 10, and 18 minus baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
Number analyzed (Participants) | 28 | 14
units on a scale
  Week 2 | -0.8 (1.7) | -0.6 (1.4)
  Week 4 | -1.0 (2.1) | -0.6 (2.1)
  Week 10 | -1.6 (3.0) | -1.1 (2.4)
  Week 18 | -2.6 (2.9) | -0.8 (1.6)

ADVERSE EVENTS:
Time Frame: From screening to last visit at 18 weeks for a total of at least 22 weeks
Arm/Group | Group 1: Experimental | Group 2: Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/14
Other Adverse Events (participants affected / at risk) | 7/28 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Experimental (N=28) | Group 2: Placebo Comparator (N=14)
urinary infection (Infections and infestations) | 7 (7) | 4 (4)

LIMITATIONS AND CAVEATS:
Limitations include a larger, longer, multi-center randomized controlled trial is warranted with the primary endpoint at 18 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02497976/SAP_000.pdf
  • Study Protocol (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02497976/Prot_001.pdf
  • Informed Consent Form (2015-07-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02497976/ICF_002.pdf